CLINICAL TRIAL: NCT07295496
Title: A Single-dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Recombinant Anti-IL-RAP Humanized Monoclonal Antibody Injection in Chinese Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetic of IBI3011
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI3011A101
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Gout Flare
Keywords: acute gout flare

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): IBI3011 placebo group
  Interventions: Drug: IBI3011 Placebo
- IBI3011 (Active Comparator): IBI3011 group
  Interventions: Drug: IBI3011

INTERVENTIONS:
Drug: IBI3011 — * Anti-IL-RAP humanised monoclonal antibody injection
  * 300 mg (2.0 mL)/vial
  * Administered in accordance with the study protocol
  * Single administration only
  Arms: IBI3011
Drug: IBI3011 Placebo — * Anti-IL-RAP humanised monoclonal antibody placebo injection
  * 300 mg (2.0 mL)/vial
  * Administered in accordance with the study protocol
  * Single administration only
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of recombinant Anti-IL-RAP humanised monoclonal antibody injection in healthy Chinese subjects (Part A) and subjects with acute gout flare (Part B)

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet all of the following Inclusion Criteria:

1. Age ≥18 years of age, male or female;
2. Body mass index (BMI) 18-26 kg/m2 (inclusive) for Part A healthy subjects and BMI 18-40 kg/m2 (inclusive) for Part B acute gout flare subjects; Part B acute gout flare subjects also needed to meet the following criteria
3. Meet ACR 2015 preliminary criteria for the classification of acute arthritis of primary gout;
4. Other inclusion criteria set by protocol

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible to attend this clinical study:

1. Difficulties in venous blood collection or a history of dizziness when encountering blood or needles;
2. Have received an experimental agent within 1 month or 5 times half-life (whichever is longer) prior;
3. Have live or attenuated vaccination in the 3 months before randomization or plan to receive that during this trial;
4. Blood donation or blood loss of more than 400 mL within 8 weeks before the screening;
5. Have a history of severe infection, severe trauma, or major surgical procedures within 6 months before the screening;
6. History of malignancy;
7. Female during pregnancy or lactation;
8. Have a history of drug abuse, drug dependence, or a positive result in a drug screen within 12 months before the screening;
9. Has a history of neuropsychiatry or any other disease/ailment that is unsuitable for this clinical trial at the discretion of the Investigator;

   Part B acute gout flare subjects also needed to exclude the following criteria:
10. Secondary gout (e.g., gout induced by chemotherapy, transplant-related gout);
11. Infection/septic arthritis, or other acute inflammatory arthritis;
12. Other exclusion criteria set by protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 12 week
  To investigate the safety characteristics.

SECONDARY OUTCOMES:
Immunogenic outcome | 12 week
  The incidence of antidrug Antibody (ADA) and/or Neutralising antibodies (NAb)
AUC | 12 Week
  Describing the Area Under Curve
Cmax | 12 Week
  Describing the Maximum Serum Concentration of Drug
CL or CL/F | 12 Week
  Describing the Clearance
V or V/F | 12 Week
  Describing the Apparent Volume of Distribution
t1/2 | 12 Week
  Describing the Half Life

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China